CLINICAL TRIAL: NCT05123807
Title: Secondary Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Recurrent Mucinous Ovarian Cancer (HI-MOC Study)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0660; NCI-2021-12842 (Other: NCI-CTRP Clinical Trials Gov Registry)
Record Dates: First submitted 2021-11-08; First posted 2021-11-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cytoreductive surgery (Other)
  Interventions: Other: Cytoreductive surgery

INTERVENTIONS:
Other: Cytoreductive surgery — (an operation to remove as much tumor tissue as possible) with hyperthermic intraperitoneal chemotherapy

SUMMARY:
The primary objective is to estimate overall survival after secondary cytoreductive surgery and HIPEC for women with recurrent primary mucinous ovarian cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

The primary objective is to estimate progression-free survival (PFS) after secondary cytoreductive surgery and HIPEC for women with recurrent primary mucinous ovarian cancer

SECONDARY OBJECTIVES:

* To estimate overall survival (OS) after secondary cytoreductive surgery and HIPEC for women with recurrent primary mucinous ovarian cancer
* To evaluate toxicity and morbidity of secondary cytoreductive surgery and HIPEC for women with recurrent primary mucinous ovarian cancer
* To estimate quality of life after secondary cytoreductive surgery and HIPEC for women with recurrent primary mucinous ovarian cancer
* To estimate what proportion of patients who preoperatively appear to be candidates for secondary cytoreductive surgery and HIPEC are found to have unresectable disease at time of surgical exploration
* To collect blood and tumor samples for biobanking to be used for exploratory endpoints

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed recurrent primary mucinous ovarian cancer
* Age ≥18 years
* ECOG performance status ≤ 2
* Prior to surgery, patients must have adequate organ and marrow function as defined below (within 30 days of registration):

  1. absolute neutrophil count >1,500/mcL
  2. platelets >100,000/mcL
  3. total bilirubin ≤ 1.5 mg/dL
  4. creatinine ≤ 1.5 mg/dL
  5. AST(SGOT)/ALT(SGPT) ≤ 3 X institutional upper limit of normal
* Patients must be > 2 weeks from prior chemotherapy or radiation therapy, except for bevacizumab treatment which requires >6 weeks
* Ability to understand and the willingness to sign a written informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of HIPEC (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Patients with mucinous tumors with pathologic confirmation of a non-gynecologic site of origin
* Patients with known active CNS metastases
* Patients with known hypersensitivity to any of the components of cisplatin
* Patients with a prior or concurrent malignancy who natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or nursing women
* Patients with peripheral neuropathy ≥ grade 2
* History of allogenic transplant
* History of prior HIPEC or intraperitoneal chemotherapy
* Known bulky extra-abdominopelvic disease
* Patients with hearing impairment/tinnitus ≥ grade 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To estimate progression-free survival (PFS) after secondary cytoreductive surgery and HIPEC for women with recurrent primary mucinous ovarian cancer | through study completion, an average of 6 years (patients will be followed for 6 years after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Shafer, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org